CLINICAL TRIAL: NCT00499759
Title: In-Hospital Individualized Prescriptive Exercise Intervention for Acute Leukemia Patients Undergoing Chemotherapy
Brief Title: Individualized Exercise Programs for Patients Receiving Chemotherapy for Newly Diagnosed Acute or Relapsed Myeloid Leukemia or Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 0526; CDR0000551972 (Other: PDQ number)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Depression; Fatigue; Leukemia; Musculoskeletal Complications; Psychosocial Effects of Cancer and Its Treatment
Keywords: fatigue; depression; psychosocial effects of cancer and its treatment; musculoskeletal complications; acute undifferentiated leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Depression; Fatigue; Leukemia; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Resting vitals — The fitness assessments will include the assessment of resting vitals including, blood pressure, heart rate, and hemoglobin saturation (pulse oximeter).
Behavioral: Body Composition — Body composition and body circumference measurements (anthropometry) will be the only assessments performed multiple times during the study to monitor possible changes in the body composition and swelling of the patients. Body composition analyses will be performed via skinfold measurements following generalized three-site skinfold equations for male and females as recommended by the ACSM, 2005 and via the utilization of a bioelectrical impedance body fat analyzer device.
Behavioral: Timed Get-up and Go test (TGUG). — The functional mobility of the subjects that will participate in the study will be assessed through the Timed Get-up and Go test (TGUG). The administration of the TGUG includes measuring a distance of 3 meters from the legs of a straight-backed armchair with a seat height of approximately 46 centimeters. The subject will be asked to sit with the back against the chair with the arms on the arm rests. When instructed to begin the test (on the command "Go"), the subject will have to stand upright then walk at a normal walking pace toward the 3 meters mark placed on the ground, turn around, return to the chair, and sit down. The stopwatch was started on the word "Go" and stopped when the subject gets back to starting position.
Behavioral: Cardiorespiratory assessment — The cardiorespiratory assessment will be performed on a recumbent cycle ergometer. Subjects will be asked to cycle at a target submaximal intensity of 60 % of their percentage of heart rate range until a RPE (Rate of Perceived Exertion) of 7 is reached on the modified Borg Scale or when the subject requests termination. The Borg modified RPE scale is a scale ranging from 0 to 11 where 0 means no exertion at all and 11 equals to an exertion of absolute maximum. The total time cycling and heart rate (HR) at the end of the test will be recorded immediately after the test is completed.
Behavioral: Handgrip evaluation — Handgrip strength will be tested using a handgrip dynamometer. Subjects will be asked to stand and hold the handgrip dynamometer in one hand lined with the forearm that will be placed beside the body. Maximum grip strength is then determined without swinging the arm and by squeezing the handgrip dynamometer as hard as possible using one brief maximal contraction with no extraneous body movement. The test will be administered three times for each hand with a one-minute rest in between trials. The best score within the three trials for each arm will be the one that will be used for analysis.
Behavioral: Dynamic muscular endurance — Subjects will be asked to squat to a 75 degree knee angle with moderate speed, pressing back against the ball at all times. This is repeated as many repetitions as it takes for the subject to report an RPE of 7 or wishes to stop. The second test is the biceps curl exercise. The biceps curls exercise test will follow a protocol developed at the Rocky Mountain Cancer Rehabilitation Institute (RMCRI), Greeley, Colorado. The protocol involves the administration of the exercise biceps curls, done with dumbbells. Subjects will be asked to perform as many repetitions as possible during an alternated biceps curl exercise using a percentage of their body weight as resistance.

SUMMARY:
RATIONALE: An individualized exercise program may be effective in lessening fatigue and depression and improving quality of life in patients undergoing chemotherapy for leukemia.

PURPOSE: This clinical trial is studying how well individualized exercise programs work in patients receiving chemotherapy for newly diagnosed acute or relapsed myeloid leukemia or lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effects, in terms of fitness and blood parameters, fatigue levels, and quality of life, of an individualized prescriptive exercise intervention in patients with newly diagnosed acute or relapsed myeloid or lymphoblastic leukemia undergoing chemotherapy.

Secondary

* Determine the feasibility of developing an exercise program for these patients.
* Assess the changes in cardiovascular endurance, muscular strength, selected blood parameters, and response of inflammatory proteins to exercise in these patients.
* Evaluate fatigue, depression, and quality of life of these patients.

OUTLINE: This is a pilot study.

Patients participate in an individualized prescriptive exercise intervention 3 to 4 times per week for 6 weeks (4 weeks in hospital, 2 weeks at home). Exercise begins concurrently with the first course (induction therapy) of chemotherapy. Each exercise session consist of 3-5 minutes of light stretching (stretching component), 5-10 minutes of cycling on the recumbent bicycle (cardiorespiratory component), 5-15 minutes of resistance training including hand dumbbells, exercise tubing, rubber bands, and fit balls (resistance training component), and 5-10 minutes of abdominal exercises (core muscles component).

Quality of life, fatigue, and depression are assessed at baseline and weekly during study intervention.

Blood samples are collected at baseline and at weeks 3 and 6 for cytokine analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute or relapsed myeloid or lymphoblastic leukemia

  * Currently receiving re-induction therapy or designated for chemotherapy treatment
* Expected hospital stay of 3-4 weeks or longer
* Participation in the study must be approved by the physician directly responsible for the patient's care while at University of North Carolina Hospitals

PATIENT CHARACTERISTICS:

* No condition that would compromise the patient's ability to participate in the exercise rehabilitation program, including any of the following:

  * Immune deficiency
  * Acute or chronic bone, joint, or muscular abnormalities
  * Acute or chronic respiratory disease
  * Cardiovascular disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Effects of an individualized prescriptive exercise intervention | 6 weeks
  All patients will participate in an individualized prescriptive exercise intervention 3 to 4 times per week (depending on the physical status of each patient during each week) for a period of 6 weeks. The exercise intervention will begin on week 1 of the study, the day after the first battery of initial assessments is concluded. Each exercise session will be divided into two bouts. One bout will be administered in the morning and the second one late in the afternoon

SECONDARY OUTCOMES:
Number of subjects experiencing fatigue, depression, and quality of life issues | 6 weeks
  The Functional Assessment of Cancer Therapy-General (FACT-G) will be administered to assess the levels of fatigue, and quality of life on weeks 2, 3 and 5 of the 6 week trial. The Center for Epidemiologic Studies Depression Scale (CES-D) will be also administered to explore the effects of exercise on depression on weeks 2, 3 and 5 of the 6 week trial.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio L. Battaglini, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States